CLINICAL TRIAL: NCT07287059
Title: Effects of Wearable Robotic and Virtual Reality-Assisted Interventions on Hand Function in Stroke Rehabilitation
Brief Title: Wearable Robotic and Virtual Reality on Hand in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Taha Ayberk Erdoğan, Physiotherapist (MSc) - Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-4330
Record Dates: First submitted 2025-11-25; First posted 2025-12-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Post-Stroke Hemiplegia
Keywords: Stroke; Soft Robotic Glove; Leap Motion Controller; Rehabilitation; Hand Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soft Robotic Glove (Experimental): Participants receive conventional Neurodevelopmental Therapy (NDT) combined with a wearable soft robotic glove (SRG) performing standard grip, tripod grip, palmar grip, and 1st-5th finger opposition tasks, 3 sessions/week for 6 weeks
  Interventions: Device: Soft Robotic Glove (SRG)
- Leap Motion Controller (Experimental): Participants receive conventional NDT combined with Leap Motion Controller integrated with the Becure HandROM and ErgoActive modules, performing LeapBall (wrist flexion/extension, abduction/adduction), Piano (finger flexion/extension), PinchPeg (precision pinch), and Hold-and-Put (palmar grasp-release) exercises, 3 sessions/week for 6 weeks.
  Interventions: Device: Leap Motion Controller (LMC)
- Control Group (Active Comparator): Participants receive NDT alone, supplemented with standard task-oriented hand exercises such as resisted wrist/hand movements, bottle grasp-release, peg transfer, and ball grasp-release activities, 3 sessions/week for 6 weeks.
  Interventions: Behavioral: Neurodevelopmental Therapy (NDT)

INTERVENTIONS:
Device: Soft Robotic Glove (SRG) — A wearable pneumatically driven soft robotic glove assisting finger flexion-extension and various grip patterns; used with NDT three sessions per week for six weeks.
  Arms: Soft Robotic Glove
Device: Leap Motion Controller (LMC) — A virtual-reality-based optical motion-tracking device combined with Becure HandROM/ErgoActive exercise modules; used with NDT three sessions per week for six weeks.
  Arms: Leap Motion Controller
Behavioral: Neurodevelopmental Therapy (NDT) — Conventional therapist-guided task-oriented upper-limb rehabilitation including resistance exercises, bottle/ball grasp-and-release, peg transfer; three sessions per week for six weeks
  Arms: Control Group

SUMMARY:
Stroke is a common neurological disorder resulting from acute focal damage to the central nervous system due to vascular events such as cerebral infarction, intracerebral hemorrhage, or subarachnoid hemorrhage. It represents one of the leading causes of mortality and long-term disability in adults, with approximately 85 % of cases being ischemic and 15 % hemorrhagic. Among survivors, up to 70 % experience upper-limb functional loss and about 40 % remain chronically impaired, particularly in wrist and hand extension due to synergy patterns and spasticity. Rehabilitation targeting upper-limb motor recovery is therefore crucial for improving activities of daily living and social participation. Technology-assisted interventions such as wearable soft robotic gloves and virtual-reality-based motion-tracking devices have recently been introduced to enhance neuroplasticity, improve voluntary movement quality, and facilitate functional independence.

This multicenter, randomized controlled clinical trial will be conducted between November 2025 and June 2026. The study will include adults aged 30-60 years with a confirmed diagnosis of post-stroke hemiplegia (ICD-10: G81) who meet the predefined inclusion criteria-including Mini-Mental State Examination > 24, Modified Ashworth Scale < 3, wrist extension > 10°, Brunnstrom stage > 3, and Fugl-Meyer Upper-Limb score > 22-will be recruited after written informed consent. Exclusion criteria include significant neglect or visual deficits, communication disorders, peripheral nerve injury, botulinum toxin injection within the previous six months, major orthopedic surgery of the affected limb, or serious systemic comorbidities. Eligible participants will be randomly assigned to one of three groups for six weeks of therapy, three sessions per week: (1) Neurodevelopmental therapy (NDT) and wearable Soft Robotic Glove (SRG); (2) NDT and Leap Motion Controller (LMC) integrated with the Becure platform (HandROM and ErgoActive modules including LeapBall, Piano, PinchPeg, and Hold-and-Put tasks); or (3) NDT-only control group performing standard task-oriented hand exercises.

Assessments will be performed at baseline and after the 18th treatment session and will include demographic data, Box-and-Block Test, Chedoke Arm and Hand Activity Inventory, surface electromyography for muscle strength, and joint-angle measurements using LMC-based Becure HandROM. The primary outcomes of this study are upper-limb functional performance and hand dexterity, while the secondary outcomes include joint range of motion, grip-pattern kinematics, and muscle strength. The findings are expected to compare and determine the effectiveness of wearable soft robotic-assisted and virtual reality-assisted interventions in post-stroke upper-limb rehabilitation, thereby guiding the evidence-based integration of advanced technologies into routine neurorehabilitation practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* Mini-Mental State Examination score > 24
* Modified Ashworth Scale score < 3
* Active wrist extension > 10°
* Brunnstrom stage > 3
* Fugl-Meyer Upper Extremity score > 22

Exclusion Criteria:

* Presence of significant unilateral neglect
* Presence of significant visual deficits
* Communication disorders that interfere with assessment or intervention
* Peripheral nerve injury affecting the upper limb
* Botulinum toxin injection to the affected upper limb within the previous six months
* History of major orthopedic surgery of the affected upper limb
* Serious systemic comorbidities
* History of epileptic seizures

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Hand Function - Chedoke Arm and Hand Activity Inventory (CAHAI) | Baseline (pre-treatment, week 0) and after 6 weeks of intervention (post-treatment, week 6)
  The Chedoke Arm and Hand Activity Inventory (CAHAI) evaluates functional bilateral task performance in individuals with post-stroke hemiplegia. It consists of 9 functional tasks scored on a 7-point scale (1 = total assistance, 7 = complete independence). Higher scores indicate better upper-limb functional performance and independence in daily activities.
Box-and-Block Test (BBT) | Baseline (pre-treatment, week 0) and after 6 weeks of intervention (post-treatment, week 6)
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. Participants move as many wooden blocks as possible from one compartment of a box to another in 60 seconds. The total number of transferred blocks is recorded; higher scores indicate better hand dexterity and motor coordination.

SECONDARY OUTCOMES:
Range-of-Motion (ROM) | Baseline (pre-treatment, week 0) and after 6 weeks of intervention (post-treatment, week 6)
  Joint kinematics of the wrist and fingers are measured using the Leap Motion Controller integrated with the Becure HandROM system. The device records angular values of flexion/extension, abduction/adduction, and radial/ulnar deviation during grasp patterns. Greater angular range indicates improved active joint mobility and motor performance.
Surface Electromyography (sEMG) | Baseline (pre-treatment, week 0) and after 6 weeks of intervention (post-treatment, week 6)
  Surface electromyography (sEMG) records electrical activity of selected upper-limb muscles during voluntary movement. Non-invasive surface electrodes are placed on the wrist and finger extensor/flexor groups to evaluate muscle activation amplitude and pattern. Increased amplitude reflects improved voluntary muscle recruitment and motor control.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Physiotherapy and Rehabilitation Department, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Background] Hung CS, Hsieh YW, Wu CY, Chen YJ, Lin KC, Chen CL, Yao KG, Liu CT, Horng YS. Hybrid Rehabilitation Therapies on Upper-Limb Function and Goal Attainment in Chronic Stroke. OTJR (Thorofare N J). 2019 Apr;39(2):116-123. doi: 10.1177/1539449218825438. Epub 2019 Mar 5. PMID 30834812
- [Background] Merletti R, Gulisashvili A, Lo Conte LR. Estimation of shape characteristics of surface muscle signal spectra from time domain data. IEEE Trans Biomed Eng. 1995 Aug;42(8):769-76. doi: 10.1109/10.398637. PMID 7642190
- [Background] Schuster C, Hahn S, Ettlin T. Objectively-assessed outcome measures: a translation and cross-cultural adaptation procedure applied to the Chedoke McMaster Arm and Hand Activity Inventory (CAHAI). BMC Med Res Methodol. 2010 Nov 29;10:106. doi: 10.1186/1471-2288-10-106. PMID 21114807
- [Background] Kolbasi EN, Ersoz Huseyinsinoglu B, Erdogan HA, Cabalar M, Bulut N, Yayla V. What are the determinants of explicit and implicit motor imagery ability in stroke patients?: a controlled study. Somatosens Mot Res. 2020 Jun;37(2):84-91. doi: 10.1080/08990220.2020.1741344. Epub 2020 Mar 31. PMID 32228207
- [Background] Oh HS, Kim EJ, Kim DY, Kim SJ. Effects of Adjuvant Mental Practice on Affected Upper Limb Function Following a Stroke: Results of Three-Dimensional Motion Analysis, Fugl-Meyer Assessment of the Upper Extremity and Motor Activity Logs. Ann Rehabil Med. 2016 Jun;40(3):401-11. doi: 10.5535/arm.2016.40.3.401. Epub 2016 Jun 29. PMID 27446776
- [Background] Proietti T, Nuckols K, Grupper J, Schwerz de Lucena D, Inirio B, Porazinski K, Wagner D, Cole T, Glover C, Mendelowitz S, Herman M, Breen J, Lin D, Walsh C. Combining soft robotics and telerehabilitation for improving motor function after stroke. Wearable Technol. 2024 Jan 26;5:e1. doi: 10.1017/wtc.2023.26. eCollection 2024. PMID 38510985
- [Background] Arman N, Oktay AB, Tarakci D, Tarakci E, Akgul YS. The validity of an objective measurement method using the Leap Motion Controller for fingers wrist, and forearm ranges of motion. Hand Surg Rehabil. 2021 Sep;40(4):394-399. doi: 10.1016/j.hansur.2021.03.007. Epub 2021 Mar 26. PMID 33781957
- [Background] Villafane JH, Taveggia G, Galeri S, Bissolotti L, Mulle C, Imperio G, Valdes K, Borboni A, Negrini S. Efficacy of Short-Term Robot-Assisted Rehabilitation in Patients With Hand Paralysis After Stroke: A Randomized Clinical Trial. Hand (N Y). 2018 Jan;13(1):95-102. doi: 10.1177/1558944717692096. Epub 2017 Feb 16. PMID 28719996
- [Background] Thimabut W, Terachinda P, Kitisomprayoonkul W. Effectiveness of a Soft Robotic Glove to Assist Hand Function in Stroke Patients: A Cross-Sectional Pilot Study. Rehabil Res Pract. 2022 Apr 25;2022:3738219. doi: 10.1155/2022/3738219. eCollection 2022. PMID 35509444
- [Background] Cortes-Perez I, Zagalaz-Anula N, Montoro-Cardenas D, Lomas-Vega R, Obrero-Gaitan E, Osuna-Perez MC. Leap Motion Controller Video Game-Based Therapy for Upper Extremity Motor Recovery in Patients with Central Nervous System Diseases. A Systematic Review with Meta-Analysis. Sensors (Basel). 2021 Mar 15;21(6):2065. doi: 10.3390/s21062065. PMID 33804247
- [Background] Crow J, Smith A. National Clinical Guideline for Stroke for the United Kingdom and Ireland: Part I - An overview of the updated recommendations. Br J Occup Ther. 2023 Oct;86(10):661-664. doi: 10.1177/03080226231188020. Epub 2023 Jul 31. No abstract available. PMID 40337193
- [Background] AVERT Trial Collaboration group. Efficacy and safety of very early mobilisation within 24 h of stroke onset (AVERT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):46-55. doi: 10.1016/S0140-6736(15)60690-0. Epub 2015 Apr 16. PMID 25892679
- [Background] Krakauer JW. Motor learning: its relevance to stroke recovery and neurorehabilitation. Curr Opin Neurol. 2006 Feb;19(1):84-90. doi: 10.1097/01.wco.0000200544.29915.cc. PMID 16415682
- [Background] Albert SJ, Kesselring J. Neurorehabilitation of stroke. J Neurol. 2012 May;259(5):817-32. doi: 10.1007/s00415-011-6247-y. Epub 2011 Oct 1. PMID 21964750
- [Background] Meschia JF, Bushnell C, Boden-Albala B, Braun LT, Bravata DM, Chaturvedi S, Creager MA, Eckel RH, Elkind MS, Fornage M, Goldstein LB, Greenberg SM, Horvath SE, Iadecola C, Jauch EC, Moore WS, Wilson JA; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Functional Genomics and Translational Biology; Council on Hypertension. Guidelines for the primary prevention of stroke: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Dec;45(12):3754-832. doi: 10.1161/STR.0000000000000046. Epub 2014 Oct 28. PMID 25355838
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265